CLINICAL TRIAL: NCT01764334
Title: A Developmental Clinical Study of Management Guided by Coronary Angiography Combined With Fractional Flow Reserve (FFR) Measurement Versus Management Guided by Coronary Angiography Alone(Standard Care) in Patients With Non-ST Elevation MI.
Brief Title: Fractional Flow Reserve Versus Angiographically Guided Management to Optimise Outcomes in Unstable Coronary Syndromes
Acronym: FAMOUS NSTEMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: British Heart Foundation (Other); Abbott Medical Devices (Industry); University of Glasgow (Other)
Responsible Party: Principal Investigator, Colin Berry, Professor Colin Berry, NHS National Waiting Times Centre Board
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: NRS-11-CA56; PG/11/55/28999 (Other Grant/Funding Number: British Heart Foundation (PG/11/55/28999))
Record Dates: First submitted 2012-12-24; First posted 2013-01-09 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: NonST Elevation Myocardial Infarction; Myocardial Infarction
Keywords: NonST elevation myocardial infarction (NSTEMI); Fractional flow reserve (FFR); Coronary angiogram; Diagnosis; Coronary revascularization; Prognosis; Health economics
MeSH Terms: conditions — Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Disease

STUDY DESIGN:
Intervention Model Description: Diagnostic intervention using fractional flow reserve
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding of FFR result
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fractional flow reserve (Active Comparator): Fractional flow reserve - guided group:
  The initial treatment decision and the coronary arteries for fractional flow reserve (FFR) measurement will be established and recorded before randomization. FFR will then be measured by the cardiologist immediately after randomization and the FFR result will used to guide treatment decisions based on a threshold of 0.80. An FFR ≤ 0.80 should result in a treatment decision for revascularization by PCI or CABG combined with optimal medical therapy and an FFR>0.80 should result in treatment with optimal medical therapy alone. Changes in treatment compared to the treatment plan prior to FFR disclosure will be recorded at the time.
  Interventions: Device: Fractional flow reserve
- Angiography-guided (Placebo Comparator): FFR is measured by but not disclosed to the clinical team. Treatment decisions are therefore guided by angiography but not by FFR. The patient and the clinical team, including the cardiologists and nurses, will be blinded to FFR. The RadiAnalyzer Xpress (St Jude Medical) will be turned away from the clinical team who will not see the pressure wire data. FFR will not be displayed on any other monitor. Quality control checks, such as assessments of equalized pressure, will be done in the usual way, by the unblinded clinical research team. These steps will be followed for all FFR measurements. Adherence to the blinding protocol, including any non-protocol FFR disclosure at any time, will be prospectively recorded and blinding procedures will be monitored with site visits.
  Interventions: Device: Fractional flow reserve

INTERVENTIONS:
Device: Fractional flow reserve — Guidewire-based coronary pressure measurement of myocardial FFR can identify obstructive coronary lesions in patients with stable coronary disease, and potentially, medically stabilized patients with recent MI. The FFR index is measured by a conventional coronary wire (0.014") with a pressure sensor on its distal tip during coronary hyperemia induced by intravenous or intracoronary adenosine. The potential diagnostic and prognostic benefit of guidewire-based coronary pressure measurement to inform the management and treatment of patients with recent acute NSTEMI will be assessed.
  Other Names: FFR; Pressure wire

SUMMARY:
Background: In patients with acute non-ST elevation myocardial infarction (NSTEMI) coronary arteriography is usually recommended however visual interpretation of the coronary angiogram is subjective. A complementary diagnostic approach involves measuring the pressure drop across a coronary stenosis (fractional flow reserve, FFR) with a pressure-sensitive guidewire.

Hypothesis: Routine FFR measurement is feasible in NSTEMI patients and has additive diagnostic, clinical and health economic utility, as compared to angiography-guided standard care.

Design: A prospective multi-center randomized controlled trial in 350 NSTEMI patients with ≥1 coronary stenosis ≥30% severity (threshold for FFR measurement). Patients will be randomized immediately after coronary angiography to the FFR-guided group or angiography-guided group (FFR measured, not disclosed). All patients will then undergo FFR measurement in all vessels with a coronary stenosis ≥30% severity. FFR will be measured in culprit and non-culprit lesions in all patients. FFR will be disclosed to guide treatment in the FFR guided-group but not disclosed in the 'angiography-guided' group. In the FFR-guided group, an FFR>0.80 will be an indication for medical therapy whereas an FFR≤0.80 will be an indication for revascularization by percutaneous coronary intervention (PCI) or coronary artery bypass surgery (CABG), as appropriate. The primary endpoint is the between-group difference in the proportion of patients allocated to medical management compared to revascularization. A key secondary composite outcome is the occurrence of cardiac death or hospitalization for myocardial infarction or heart failure. Other secondary outcomes include quality of life, hospitalization for unstable angina, coronary revascularization or stroke, and healthcare costs. Exploratory analyses will also assess the relationships between FFR and angiographic lesion characteristics (severity, culprit status). The minimum and average follow-up periods for the primary analysis are 6 and 18 months respectively. A secondary analysis with longer term follow-up (minimum 3 years) is planned. Screen failures who gave informed consent will be entered into a registry.

Importance: Our developmental clinical trial will address the feasibility of FFR measurement in NSTEMI and the influence of FFR disclosure on treatment decisions and health and economic outcomes.

DETAILED DESCRIPTION:
Background

Acute non-ST elevation myocardial infarction (NSTEMI) is the commonest form of acute coronary syndrome (ACS) and a leading global cause of premature morbidity and mortality. A coronary angiogram is recommended in intermediate-high risk NSTEMI patients to detect obstructive coronary artery disease (CAD) and so identify patients who may benefit from coronary revascularization. In ACS patients, stress testing before invasive management is not recommended and so functional information on ischemia is usually not available. Therefore, usual care is based on visual interpretation of coronary disease severity revealed by the angiogram and treatment decisions include medical therapy, percutaneous coronary intervention (PCI) or coronary artery bypass surgery (CABG). Since visual assessment of the angiogram may be inaccurate, judgements made by cardiologists in every day practice are subjective, potentially leading to misdiagnosis and incorrect treatment decisions.

Recent studies (DEFER, FAME, FAME II) in patients with stable coronary artery disease (CAD) have presented a new approach to the diagnostic management of CAD. Fractional flow reserve (FFR) is an index of the physiological significance of a coronary stenosis and is defined as the ratio of maximal blood flow in a stenotic artery to normal maximal flow. An FFR ≤0.80 is an evidence-based physiological threshold that correlates with the presence of inducible ischemia on non-invasive testing. Alternatively, an FFR >0.80 indicates that patients can be managed safely with medical therapy. DEFER and FAME highlighted the benefits of FFR measurement in stable CAD to more accurately identify flow-limiting stenoses and guide PCI leading to improved outcomes and reduced costs compared to angiography alone. In FAME 2, compared to optimal medical therapy alone, PCI combined with optimal medical therapy reduced the likelihood of urgent revascularization in patients with stable symptoms and functionally significant coronary disease. Overall, FFR measurement can identify and exclude obstructive coronary artery disease with high diagnostic accuracy, including in patients with prior MI.

FFR measurement in unstable coronary artery disease

There is some uncertainty over the validity of FFR when measured in patients with recent MI. FFR measurement requires maximal coronary hyperemia which theoretically may be less readily achieved in patients with recent MI, potentially, because of microvascular injury.

The results of several recent studies support the notion that FFR measurements are valid in medically stabilized MI patients. First, Ntalianis et al measured FFR in 112 non-culprit coronary lesions repeatedly (average interval 35±4 days) in 101 patients with recent MI and found similar FFR values at each time-point. In one other study, FFR correctly identified inducible ischemia on SPECT in 57 patients >6 days after MI and in one other study of 124 ACS patients, deferring revascularization in lesions with an FFR ≥ 0.75 was safe during longer term follow-up. In hospitalized patients with recent MI and angiographic intermediate coronary lesions, FFR-guided management reduced in-hospital costs compared to deferred management with revascularization guided by myocardial stress perfusion scintigraphy. Finally, nearly one third of the patients randomized in FAME had a history of medically stabilized unstable angina or NSTEMI five or more days from randomization. The FAME investigators performed a post-hoc analysis of these patients and found a similar risk reduction for major adverse cardiovascular events in the FFR group compared to the angiography-guided group leading them to conclude that the benefit of using FFR to guide PCI in multivessel disease may not differ between patients with unstable vs. stable coronary disease. The FAME investigators concluded that their post hoc analysis could not prove equivalence of effects between subgroups since FAME was neither designed nor powered to do so.

Therefore, the potential diagnostic, prognostic and health economic impact of FFR measurement to inform the management of unselected patients with recent (i.e. < 5 days) medically stabilized NSTEMI has not been established.

Specific uncertainties with angiography-guided treatment decisions in NSTEMI.

First, treatment decisions for non-obstructive (FFR>0.80) culprit CAD lack an evidence base to guide management. On the one hand, a stent which covers a ruptured coronary plaque might reduce the risks of recurrent thrombosis. On the other hand, optimal medical therapy with dual anti-platelet drugs and high dose statins might suffice and unnecessary stenting can be harmful (e.g. stent thrombosis). Second, in NSTEMI patients with multivessel coronary disease, evidence is lacking as to whether non-culprit obstructive lesions should undergo revascularization or not. A post-hoc analyses of the contemporary large scale Acute Catheterization and Urgent Intervention Triage Strategy (ACUITY) trial found that incomplete coronary revascularization was a multivariable predictor of major adverse cardiac events at 1 year and the risk was related to the number of non-revascularized lesions. A post hoc analysis of NSTEMI patients treated during usual care has found that FFR disclosure does influence cardiologists' treatment decisions leading to improved diagnostic efficiency compared angiography-guided decisions. Third, uncertainties remain about whether maximal coronary hyperemia can be achieved in patients with recent MI using the standard dose of adenosine (140 micrograms/kg/min) or whether higher doses of adenosine (170 - 210 micrograms/kg/min) might be needed. This question is relevant since sub-maximal coronary vasodilatation could be associated with a falsely elevated FFR value which in turn could result in an inappropriate decision in favor of medical therapy rather than revascularization.

Rationale for a trial of FFR-guided management vs. angiography alone in NSTEMI.

FFR measurement is not a current standard of care in NSTEMI patients. Therefore, in our study, FFR will be measured but not disclosed in the angiography-guided control group. Second, FFR values and their relationships with clinical outcomes may differ in patients with unstable coronary disease compared to patients with stable coronary disease. In our trial, FFR will be measured in all patients including in the angiography-guided control group (175 patients) in whom FFR will be measured but not disclosed to the clinical team responsible for the patient. Since patients will be followed-up for clinical events, the relationships (and ROC values) between FFR and health outcomes (composite cardiovascular events) will be prospectively evaluated.

Third, since stress testing is not appropriate in acute MI patients, FFR-guided management could obviate the need for 'deferred' management. Fourth, FFR has the potential to guide the decision for or against revascularization of culprit and non-culprit lesions. Since there are no data to support stenting in lesions which are not functionally significant, the investigators propose that the treatment decisions are consistently guided by the FFR values in both culprit and non-culprit arteries using the established FFR threshold of 0.80 for revascularization. Non-flow limiting lesions (FFR>0.80) would be treated with optimal medical therapy and flow-limiting lesions (FFR≤0.80) should revascularized by PCI or CABG. Fifth, when stenting is performed, the post-stent FFR can be used to ensure that an optimal stent result is achieved i.e. an FFR >0.9 in both the culprit and non-culprit lesions treated by PCI.

Study Hypothesis

Routine FFR measurement is feasible in NSTEMI patients and has additive diagnostic, clinical and health economic utility, as compared to current standards of care based on visual assessment of the angiogram.

Methodology

Overall aim: To generate evidence that will permit (or not) the development of new diagnostic and disease management strategies which will accurately and efficiently distinguish between flow limiting and non-flow limiting coronary stenoses, a major challenge in current revascularization strategies in patients with recent MI directed by angiography alone.

Primary Aims:

1) To determine if the treatment and outcomes of NSTEMI patients whose management is guided by FFR disclosure differ compared to patients whose treatment is guided by visual interpretation of the angiogram alone (FFR measured, not disclosed).

Secondary Aims:

1. To determine the feasibility and safety of routine coronary guidewire-based FFR measurement in NSTEMI,
2. To determine the level of agreement between functional (FFR) and visual assessments of coronary disease severity in NSTEMI patients,
3. To assess the proportion of patients with a clinical response to adenosine (initial dose of 140 µg/kg/min, maximum dose 210 µg/kg/min), as revealed by typical changes in heart rate and blood pressure and the occurrence of patient symptoms,
4. To determine the relationships between FFR values during the baseline procedure (and receiver operating characteristic) and cardiac events during follow-up in all patients,
5. To provide preliminary data on whether FFR-guided management is associated with improved health outcomes and quality of life in the longer term compared to angiography-guided treatment decisions,
6. To perform a health-economic analysis.

Standard care of NSTEMI patients in the UK National Health Service

The participating hospitals adhere to current guidelines for optimal medical therapy and optimal revascularization. A left main stenosis of >50% and an epicardial coronary stenosis >70% are usually taken to be obstructive lesions for which revascularization should be considered. In usual care, FFR is normally measured in a minority of patients (<10% of patients overall) and is not standard care. Patients who may be candidates for CABG will be discussed at the Multidisciplinary Heart Team meeting in each center. If staged PCI is clinically indicated then all procedures should take place during the index hospitalization.

Setting and Design

A prospective randomized controlled trial will be conducted in up to 6 UK centers including 3 academic cardiothoracic centers and 3 non-academic regional hospitals.

Study population

The investigators estimate 1400 consecutive NSTEMI patients with known or suspected Type 1 MI will be screened before coronary angiography. The inclusion and exclusion criteria are listed below. Patients who have given informed consent but were not randomized will be included in a follow-up registry.

Catheter laboratory study protocol

Once the coronary angiogram has been obtained, the cardiologist will assess whether or not the patient is eligible based on angiographic criteria to continue in the study and be randomized. If this is the case, randomization should take place immediately in the catheter laboratory. All eligible patients will be included wherever possible to minimize selection bias.

The main angiographic inclusion criterion is the presence of one or more non-critical coronary stenoses ≥30% severity which are (1) amenable to revascularization, (2) associated with normal coronary blood flow (TIMI grade III) and (3) in the opinion of the attending cardiologist FFR measurement is feasible and may have diagnostic value. Although an epicardial coronary stenosis of 70% is usually accepted as a threshold for revascularization, a minimum stenosis severity of 30% is adopted for FFR measurement in our study because stenosis severity may be visually underestimated. Inclusion of a stenosis >90% severity is permissible provided the cardiologist believes FFR has the potential to influence the treatment decision based on coronary and patient characteristics. Left main stem disease is included and the upper limit for stenosis severity is 80%. The pressure wire (Certus, St Jude Medical, Uppsala) will be used to provide an FFR value across all coronary narrowings ≥30% severity as appropriate.

Randomization

Once the coronary angiogram has been acquired, the cardiologist will then confirm whether or not the patient is eligible for randomization. In this case, before randomization the cardiologist will initially state the treatment plan based on the available clinical information including the angiogram. The treatment plan will then be recorded by the research team. Next, randomization will then follow-on immediately using a web-based computer randomization tool provided by the independent Clinical Trials Unit. Ineligible patients will be entered into a registry.

FFR informed group: FFR will be measured by the cardiologist immediately after randomization and the FFR result will used to guide treatment decisions based on a threshold of 0.80. An FFR ≤ 0.80 should result in a treatment decision for revascularization by PCI or CABG combined with optimal medical therapy and an FFR>0.80 should result in treatment with optimal medical therapy alone. Changes in treatment compared to the treatment plan prior to FFR disclosure will be recorded at the time.

Angiography-guided group and blinding: The patient and the clinical team responsible for the patient, including the interventional cardiologists and nurses, will be blinded to FFR. The RadiAnalyzer Xpress (St Jude Medical, Uppsala) will be turned away such that it is impossible for the clinical team to see the data which will be collected by the research team. The pressure wire recording will not be displayed on any other monitor in the catheter laboratory. Quality control checks, such as assessments of equalized pressure recordings and verification of hemodynamic changes with intravenous adenosine, will be conducted in the usual way, with the guidance of the unblinded clinical research team. These steps will be followed for all FFR measurements. Adherence to the blinding protocol, including any non-protocol disclosure of FFR at any time, will be prospectively recorded and blinding procedures will be monitored with site visits.

ELIGIBILITY:
Inclusion Criteria:

1. NSTEMI with an elevated troponin (> upper limit of normal for local reference range) with at least one CAD risk factor (e.g. diabetes, age > 65 years, prior CAD, prior peripheral vascular disease, hypertension, hyperlipidaemia, family history of CAD).
2. At least one coronary lesion ≥ 30% stenosis severity.
3. Invasive management scheduled within 10 days of admission and ideally performed within 72 h of admission or a history of recurrent ischemic symptoms within 5 days.

Exclusion Criteria:

1. On-going ischemic symptoms (i.e. chest pain) not controlled by medical therapy.
2. Cardiogenic shock or hemodynamic instability.
3. Angiographic exclusion: highly tortuous or calcified arteries, left main stenosis >80% angiographically (i.e. consistent with severe left main disease).
4. Life expectancy of < 1 year.
5. MI with persistent ST elevation.
6. Intolerance to anti-platelet drugs.
7. Unsuitable for either PCI or CABG on clinical or angiographic grounds.
8. Coronary artery disease < 30% reference vessel diameter.
9. Absence of a non-flow limiting coronary stenosis ≥30%.
10. Non-coronary cardiac surgery (e.g. concomitant valve repair or replacement).
11. Inability to give informed consent.
12. Age < 18 years (no upper age limit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2011-10; Primary Completion 2014-06 (Actual); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
The between-group difference in the proportion of patients allocated to medical management compared to revascularization. | Baseline: the treatment decision will be made by the clinical team in the cardiac catheter laboratory during the index procedure or shortly afterwards during the index hospitalization when a multidisciplinary heart team review is indicated.
  The between-group difference in the proportion of patients allocated to medical management compared to coronary revascularization by percutaneous coronary intervention (PCI) or coronary artery bypass surgery (CABG).

SECONDARY OUTCOMES:
The safety and feasibility of routine FFR measurement in patients with recent NSTEMI. | Post randomization index procedure at baseline.
  The safety of FFR measurement will be assessed by the occurrence of procedure-related adverse events including procedure-related myocardial infarction (Type 4a), coronary guidewire dissection, procedure duration and contrast nephropathy.
  The feasibility of FFR measurement will be assessed by (1) the proportion of patients who have given informed consent and who are deemed eligible for a pressure wire study and (2) the proportion of patients in whom a pressure wire study is achieved based on the number of patients in whom a pressure wire study was attempted.
The % rate of discordance between an FFR <= or >0.80 and coronary stenosis severity (stenosis > or <70% of reference vessel diameter (50% for left main) assessed visually). | Baseline: Visual assessment of the angiogram before randomization, index procedure
  The severity of coronary artery lesion(s) revealed by diagnostic coronary angiography will be visually assessed by the attending interventional cardiologist in the cardiac catheter laboratory in line with usual care. The assessment will be made and documented before randomization.
  FFR will be measured during diagnostic coronary angiography and before PCI.
Major adverse cardiac events are defined as cardiac death or hospitalization for myocardial infarction (MI) or heart failure. | Post-randomization (any time including the index procedure through follow-up), expected average follow-up of 18 months (minimum follow-up 6 months).
  Major adverse cardiovascular events are defined as cardiovascular death or hospitalization for MI, heart failure, stroke or transient ischemic attack. Information on hospitalizations for other adverse events (i.e. unstable angina, renal failure, PCI, CABG) will be prospectively recorded. Receiver-operating-characteristics will be calculated for FFR in all patients and subsequent adverse events. The endpoints will be assessed during the study until the final randomized patient has completed a minimum of 6 months follow-up. The 3-year event rates will also be assessed.
Health economics | Post-randomization (including the index procedure through longer term mean follow-up of 18 months (minimum follow-up 6 months).
  Health-care costs (including revascularization procedures, stents, bed days etc) will be prospectively recorded for the index and any subsequent hospitalizations.
Quality of life | Baseline through longer term follow-up (average follow-up 18 months, minimum follow-up 6 months)
  Quality of life (EurQoL, EQ-5D-5L) assessed at 6 monthly intervals until the last randomized patient has completed a minimum of 6 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Berry, MD PhD, Principal Investigator — University of Glasgow; Robert Henderson, MD FRCP, Study Chair — Nottingham University Hospitals, Nottingham, UK; Ian Ford, PhD, Study Director — Robertson Centre for Biostatistics - University of Glasgow; Andrew Briggs, PhD, Study Director — Health Economics and Health Technology Assessment, University of Glasgow
Locations (6):
- United Kingdom (6):
  - Golden Jubilee National Hospital, Clydebank, Dunbartonshire
  - Royal Blackburn Hospital, Blackburn, East Lancashire
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Hairmyres Hospital, East Kilbride, Lanarkshire
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - City Hospitals Sunderland NHS Foundation, Sunderland, Tyne and Wear

IPD SHARING:
Plan to Share IPD: Yes
Data sharing for the purposes of collaborative research is possible pending regulatory approval and institutional data sharing agreements.

REFERENCES:
- [Background] Hamm CW, Bassand JP, Agewall S, Bax J, Boersma E, Bueno H, Caso P, Dudek D, Gielen S, Huber K, Ohman M, Petrie MC, Sonntag F, Uva MS, Storey RF, Wijns W, Zahger D; ESC Committee for Practice Guidelines. ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: The Task Force for the management of acute coronary syndromes (ACS) in patients presenting without persistent ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2011 Dec;32(23):2999-3054. doi: 10.1093/eurheartj/ehr236. Epub 2011 Aug 26. No abstract available. PMID 21873419
- [Background] Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS); European Association for Percutaneous Cardiovascular Interventions (EAPCI); Wijns W, Kolh P, Danchin N, Di Mario C, Falk V, Folliguet T, Garg S, Huber K, James S, Knuuti J, Lopez-Sendon J, Marco J, Menicanti L, Ostojic M, Piepoli MF, Pirlet C, Pomar JL, Reifart N, Ribichini FL, Schalij MJ, Sergeant P, Serruys PW, Silber S, Sousa Uva M, Taggart D. Guidelines on myocardial revascularization. Eur Heart J. 2010 Oct;31(20):2501-55. doi: 10.1093/eurheartj/ehq277. Epub 2010 Aug 29. No abstract available. PMID 20802248
- [Background] Selby JV, Fireman BH, Lundstrom RJ, Swain BE, Truman AF, Wong CC, Froelicher ES, Barron HV, Hlatky MA. Variation among hospitals in coronary-angiography practices and outcomes after myocardial infarction in a large health maintenance organization. N Engl J Med. 1996 Dec 19;335(25):1888-96. doi: 10.1056/NEJM199612193352506. PMID 8948565
- [Background] White CW, Wright CB, Doty DB, Hiratza LF, Eastham CL, Harrison DG, Marcus ML. Does visual interpretation of the coronary arteriogram predict the physiologic importance of a coronary stenosis? N Engl J Med. 1984 Mar 29;310(13):819-24. doi: 10.1056/NEJM198403293101304. PMID 6700670
- [Background] Botman KJ, Pijls NH, Bech JW, Aarnoudse W, Peels K, van Straten B, Penn O, Michels HR, Bonnier H, Koolen JJ. Percutaneous coronary intervention or bypass surgery in multivessel disease? A tailored approach based on coronary pressure measurement. Catheter Cardiovasc Interv. 2004 Oct;63(2):184-91. doi: 10.1002/ccd.20175. PMID 15390344
- [Background] Pijls NH, van Schaardenburgh P, Manoharan G, Boersma E, Bech JW, van't Veer M, Bar F, Hoorntje J, Koolen J, Wijns W, de Bruyne B. Percutaneous coronary intervention of functionally nonsignificant stenosis: 5-year follow-up of the DEFER Study. J Am Coll Cardiol. 2007 May 29;49(21):2105-11. doi: 10.1016/j.jacc.2007.01.087. Epub 2007 May 17. PMID 17531660
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] De Bruyne B, Pijls NH, Kalesan B, Barbato E, Tonino PA, Piroth Z, Jagic N, Mobius-Winkler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd KG, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Juni P, Fearon WF; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI versus medical therapy in stable coronary disease. N Engl J Med. 2012 Sep 13;367(11):991-1001. doi: 10.1056/NEJMoa1205361. Epub 2012 Aug 27. PMID 22924638
- [Background] Fearon WF, Bornschein B, Tonino PA, Gothe RM, Bruyne BD, Pijls NH, Siebert U; Fractional Flow Reserve Versus Angiography for Multivessel Evaluation (FAME) Study Investigators. Economic evaluation of fractional flow reserve-guided percutaneous coronary intervention in patients with multivessel disease. Circulation. 2010 Dec 14;122(24):2545-50. doi: 10.1161/CIRCULATIONAHA.109.925396. Epub 2010 Nov 29. PMID 21126973
- [Background] Bech GJ, Droste H, Pijls NH, De Bruyne B, Bonnier JJ, Michels HR, Peels KH, Koolen JJ. Value of fractional flow reserve in making decisions about bypass surgery for equivocal left main coronary artery disease. Heart. 2001 Nov;86(5):547-52. doi: 10.1136/heart.86.5.547. PMID 11602550
- [Background] De Bruyne B, Pijls NH, Bartunek J, Kulecki K, Bech JW, De Winter H, Van Crombrugge P, Heyndrickx GR, Wijns W. Fractional flow reserve in patients with prior myocardial infarction. Circulation. 2001 Jul 10;104(2):157-62. doi: 10.1161/01.cir.104.2.157. PMID 11447079
- [Background] Tonino PA, Fearon WF, De Bruyne B, Oldroyd KG, Leesar MA, Ver Lee PN, Maccarthy PA, Van't Veer M, Pijls NH. Angiographic versus functional severity of coronary artery stenoses in the FAME study fractional flow reserve versus angiography in multivessel evaluation. J Am Coll Cardiol. 2010 Jun 22;55(25):2816-21. doi: 10.1016/j.jacc.2009.11.096. PMID 20579537
- [Background] Uren NG, Crake T, Lefroy DC, de Silva R, Davies GJ, Maseri A. Reduced coronary vasodilator function in infarcted and normal myocardium after myocardial infarction. N Engl J Med. 1994 Jul 28;331(4):222-7. doi: 10.1056/NEJM199407283310402. PMID 7832835
- [Background] Ntalianis A, Sels JW, Davidavicius G, Tanaka N, Muller O, Trana C, Barbato E, Hamilos M, Mangiacapra F, Heyndrickx GR, Wijns W, Pijls NH, De Bruyne B. Fractional flow reserve for the assessment of nonculprit coronary artery stenoses in patients with acute myocardial infarction. JACC Cardiovasc Interv. 2010 Dec;3(12):1274-81. doi: 10.1016/j.jcin.2010.08.025. PMID 21232721
- [Background] Potvin JM, Rodes-Cabau J, Bertrand OF, Gleeton O, Nguyen CN, Barbeau G, Proulx G, De Larochelliere R, Dery JP, Batalla N, Dana A, Facta A, Roy L. Usefulness of fractional flow reserve measurements to defer revascularization in patients with stable or unstable angina pectoris, non-ST-elevation and ST-elevation acute myocardial infarction, or atypical chest pain. Am J Cardiol. 2006 Aug 1;98(3):289-97. doi: 10.1016/j.amjcard.2006.02.032. Epub 2006 Jun 6. PMID 16860011
- [Background] Leesar MA, Abdul-Baki T, Akkus NI, Sharma A, Kannan T, Bolli R. Use of fractional flow reserve versus stress perfusion scintigraphy after unstable angina. Effect on duration of hospitalization, cost, procedural characteristics, and clinical outcome. J Am Coll Cardiol. 2003 Apr 2;41(7):1115-21. doi: 10.1016/s0735-1097(03)00057-3. PMID 12679210
- [Background] Sels JW, Tonino PA, Siebert U, Fearon WF, Van't Veer M, De Bruyne B, Pijls NH. Fractional flow reserve in unstable angina and non-ST-segment elevation myocardial infarction experience from the FAME (Fractional flow reserve versus Angiography for Multivessel Evaluation) study. JACC Cardiovasc Interv. 2011 Nov;4(11):1183-9. doi: 10.1016/j.jcin.2011.08.008. PMID 22115657
- [Background] Rosner GF, Kirtane AJ, Genereux P, Lansky AJ, Cristea E, Gersh BJ, Weisz G, Parise H, Fahy M, Mehran R, Stone GW. Impact of the presence and extent of incomplete angiographic revascularization after percutaneous coronary intervention in acute coronary syndromes: the Acute Catheterization and Urgent Intervention Triage Strategy (ACUITY) trial. Circulation. 2012 May 29;125(21):2613-20. doi: 10.1161/CIRCULATIONAHA.111.069237. Epub 2012 May 1. PMID 22550156
- [Background] Carrick D, Behan M, Foo F, Christie J, Hillis WS, Norrie J, Oldroyd KG, Berry C. Usefulness of fractional flow reserve to improve diagnostic efficiency in patients with non-ST elevation myocardial infarction. Am J Cardiol. 2013 Jan 1;111(1):45-50. doi: 10.1016/j.amjcard.2012.08.046. Epub 2012 Oct 2. PMID 23040601
- [Background] Balachandran KP, Berry C, Norrie J, Vallance BD, Malekianpour M, Gilbert TJ, Pell AC, Oldroyd KG. Relation between coronary pressure derived collateral flow, myocardial perfusion grade, and outcome in left ventricular function after rescue percutaneous coronary intervention. Heart. 2004 Dec;90(12):1450-4. doi: 10.1136/hrt.2003.023606. PMID 15547027
- [Background] Berry C, Layland J, Sood A, Curzen NP, Balachandran KP, Das R, Junejo S, Henderson RA, Briggs AH, Ford I, Oldroyd KG. Fractional flow reserve versus angiography in guiding management to optimize outcomes in non-ST-elevation myocardial infarction (FAMOUS-NSTEMI): rationale and design of a randomized controlled clinical trial. Am Heart J. 2013 Oct;166(4):662-668.e3. doi: 10.1016/j.ahj.2013.07.011. Epub 2013 Aug 27. PMID 24093845
- [Background] Layland J, Berry C. Intracoronary Adenosine for Maximal Hyperemia: Less Is More...More or Less? JACC Cardiovasc Interv. 2015 Sep;8(11):1431-1432. doi: 10.1016/j.jcin.2015.04.027. No abstract available. PMID 26404194
- [Background] Layland J, Nerlekar N, Palmer S, Berry C, Oldroyd K. Invasive assessment of the coronary microcirculation in the catheter laboratory. Int J Cardiol. 2015 Nov 15;199:141-9. doi: 10.1016/j.ijcard.2015.05.190. Epub 2015 Jul 8. PMID 26197399
- [Background] Layland J, Carrick D, McEntegart M, Ahmed N, Payne A, McClure J, Sood A, McGeoch R, MacIsaac A, Whitbourn R, Wilson A, Oldroyd K, Berry C. Vasodilatory capacity of the coronary microcirculation is preserved in selected patients with non-ST-segment-elevation myocardial infarction. Circ Cardiovasc Interv. 2013 Jun;6(3):231-6. doi: 10.1161/CIRCINTERVENTIONS.112.000180. Epub 2013 Jun 11. PMID 23756697
- [Result] Layland J, Rauhalammi S, Lee MM, Ahmed N, Carberry J, Teng Yue May V, Watkins S, McComb C, Mangion K, McClure JD, Carrick D, O'Donnell A, Sood A, McEntegart M, Oldroyd KG, Radjenovic A, Berry C. Diagnostic Accuracy of 3.0-T Magnetic Resonance T1 and T2 Mapping and T2-Weighted Dark-Blood Imaging for the Infarct-Related Coronary Artery in Non-ST-Segment Elevation Myocardial Infarction. J Am Heart Assoc. 2017 Mar 31;6(4):e004759. doi: 10.1161/JAHA.116.004759. PMID 28364045
- [Result] Nam J, Briggs A, Layland J, Oldroyd KG, Curzen N, Sood A, Balachandran K, Das R, Junejo S, Eteiba H, Petrie MC, Lindsay M, Watkins S, Corbett S, O'Rourke B, O'Donnell A, Stewart A, Hannah A, McConnachie A, Henderson R, Berry C. Fractional flow reserve (FFR) versus angiography in guiding management to optimise outcomes in non-ST segment elevation myocardial infarction (FAMOUS-NSTEMI) developmental trial: cost-effectiveness using a mixed trial- and model-based methods. Cost Eff Resour Alloc. 2015 Nov 14;13:19. doi: 10.1186/s12962-015-0045-9. eCollection 2015. PMID 26578850
- [Result] Ahmed N, Layland J, Carrick D, Petrie MC, McEntegart M, Eteiba H, Hood S, Lindsay M, Watkins S, Davie A, Mahrous A, Carberry J, Teng V, McConnachie A, Curzen N, Oldroyd KG, Berry C. Safety of guidewire-based measurement of fractional flow reserve and the index of microvascular resistance using intravenous adenosine in patients with acute or recent myocardial infarction. Int J Cardiol. 2016 Jan 1;202:305-10. doi: 10.1016/j.ijcard.2015.09.014. Epub 2015 Sep 18. PMID 26418191
- [Result] Layland J, Rauhalammi S, Watkins S, Ahmed N, McClure J, Lee MM, Carrick D, O'Donnell A, Sood A, Petrie MC, May VT, Eteiba H, Lindsay M, McEntegart M, Oldroyd KG, Radjenovic A, Berry C. Assessment of Fractional Flow Reserve in Patients With Recent Non-ST-Segment-Elevation Myocardial Infarction: Comparative Study With 3-T Stress Perfusion Cardiac Magnetic Resonance Imaging. Circ Cardiovasc Interv. 2015 Aug;8(8):e002207. doi: 10.1161/CIRCINTERVENTIONS.114.002207. PMID 26253733
- [Result] Berry C, Corcoran D, Hennigan B, Watkins S, Layland J, Oldroyd KG. Fractional flow reserve-guided management in stable coronary disease and acute myocardial infarction: recent developments. Eur Heart J. 2015 Dec 1;36(45):3155-64. doi: 10.1093/eurheartj/ehv206. Epub 2015 Jun 2. PMID 26038588
- [Result] Layland J, Oldroyd KG, Curzen N, Sood A, Balachandran K, Das R, Junejo S, Ahmed N, Lee MM, Shaukat A, O'Donnell A, Nam J, Briggs A, Henderson R, McConnachie A, Berry C; FAMOUS-NSTEMI investigators. Fractional flow reserve vs. angiography in guiding management to optimize outcomes in non-ST-segment elevation myocardial infarction: the British Heart Foundation FAMOUS-NSTEMI randomized trial. Eur Heart J. 2015 Jan 7;36(2):100-11. doi: 10.1093/eurheartj/ehu338. Epub 2014 Sep 1. PMID 25179764
- [Result] Layland J, Carrick D, Lee M, Oldroyd K, Berry C. Adenosine: physiology, pharmacology, and clinical applications. JACC Cardiovasc Interv. 2014 Jun;7(6):581-91. doi: 10.1016/j.jcin.2014.02.009. Epub 2014 May 14. PMID 24835328
- See also: Institute of Cardiovascular and Medical Sciences, University of Glasgow — http://www.gla.ac.uk/researchinstitutes/icams/
- See also: British Heart Foundation — https://www.bhf.org.uk/research